CLINICAL TRIAL: NCT01580436
Title: Prospective, Randomized Evaluation of Prophylactic Tricuspid Valve Annuloplasty in Patients Undergoing Mitral Valve Surgery
Brief Title: Prophylactic Tricuspid Valve Annuloplasty in Patients Undergoing Mitral Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, MD PhD, Professor Cardiovascular Physiology, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVP Study
Record Dates: First submitted 2011-10-18; First posted 2012-04-19 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Tricuspid Valve Insufficiency
Keywords: Tricuspid Valve Insufficiency; Cardiac Valve Annuloplasty; Outcome Assessment (Health Care)
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tricuspid Valve Annuloplasty (Experimental): Patients, undergoing mitral valve surgery with no significant tricuspid valve regurgitation despite tricuspid annular dilation, randomized to concomitant tricuspid valve annuloplasty.
  Interventions: Procedure: Tricuspid Valve Annuloplasty
- Conservative arm (No Intervention): Patients, undergoing mitral valve surgery with no significant tricuspid valve regurgitation despite tricuspid annular dilation, randomized to mitral valve surgery without concomitant tricuspid valve annuloplasty.

INTERVENTIONS:
Procedure: Tricuspid Valve Annuloplasty — Concomitant Tricuspid Valve Annuloplasty in patients undergoing mitral valve surgery
  Arms: Tricuspid Valve Annuloplasty

SUMMARY:
De novo or progressive tricuspid regurgitation (TR) is not uncommonly observed following mitral valve surgery and associated with worse outcome. Hence, concomitant tricuspid valve annuloplasty (TVP) has been recommended for patients undergoing mitral valve surgery when tricuspid annular dilatation is present even in absence of significant TR. However, whether such a strategy of "prophylactic TVP" results in improved outcomes has not been shown to date by a prospective randomized study. The investigators goal is therefore to initiate such a study and evaluate the effect of concomitant TVP on mid- and long-term outcome in patients scheduled for mitral valve surgery and tricuspid annular dilatation but <2+ TR.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for mitral valve surgery
* Tricuspid Annular diameter > 40mm or >21mm/m²

Exclusion Criteria:

* Tricuspid Regurgitation more than 2+
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
combination of all-cause mortality or heart failure hospitalisation | at 12 months post-surgery

SECONDARY OUTCOMES:
RV function & geometry | 3, 6, 12 and 18 months
  volumes and ejection fraction Assessed by cardiac ultrasound and MRI
Quality of Life | 6, 12 and 18 months
  Change at follow-up, measured by SF-36 & Minnesota Living with Heart Failure scale.
Duration of Hospital and ICU stay | postoperative phase
All-Cause Mortality | at 3, 6, 12 and 18 months post-surgery
Hospitalization for Heart Failure | at 3, 6, 12 and 18 months post-surgery
progressive TR > 2+ post-surgery | 3, 6, 12 and 18 months
cardiovascular mortality | at 3, 6, 12 and 18 months post-surgery
Exercise Tolerance | 6, 12 and 18 months
  Change at follow-up, by 6-minute walking distance and maximal exercise cyclo-ergometry (maximal aerobic capacity)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg (General Hospital Genk), Genk, Belgium